CLINICAL TRIAL: NCT04462367
Title: Clinical and Laboratory Predictors of COVID-19 Progression and Maternal and Perinatal Outcomes in Infected Pregnant and Postpartum Women in Six Reference Centers in the Northeast of Brazil
Brief Title: Northeast COVID-19 and Pregnancy Study Group
Acronym: NCOVIP
Status: Active, not recruiting | Type: Observational
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Leila Katz, Principal Investigator, Instituto Materno Infantil Prof. Fernando Figueira
Other Study IDs: NCOVIP
Record Dates: First submitted 2020-06-23; First posted 2020-07-08 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: COVID19; Coronavirus Infection; Pregnancy Disease; Severe Acute Respiratory Syndrome
Keywords: coronavirus; COVID-19; coronavirus infection; severe acute respiratory syndrome; coronavirus 2; SRAS-CoV-2; pregnancy; maternal mortality; perinatal mortality
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome; Maternal Death; Perinatal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective and retrospective cohort study. The objective will to determine the frequency of COVID-19 in pregnant and postpartum women hospitalized with flu syndrome, to evaluate clinical and laboratory predictors of COVID-19 progression and to determine the factors associated with adverse maternal and perinatal outcomes in healthcare centers in two states of Northeast Brazil.The study will be conducted including pregnant and postpartum women with clinical or laboratorial diagnosis of COVID-19, admitted in six healthcare centers in the Northeast of Brazil. All pregnant and postpartum women with clinical and/or diagnosis of COVID-19, attended in prenatal care, in emergency (maternity triage), high-risk pregnancy ward, obstetric intensive care unit and rooming-in ward will be included. The data will be collected in specific forms. The exams will be carried out by trained professionals within each institution.

DETAILED DESCRIPTION:
General Objective: To determine the frequency of COVID-19 in pregnant and postpartum women admitted with flu syndrome, to evaluate the clinical and laboratory predictors of COVID-19 progression and to identify the factors associated with adverse maternal and perinatal / neonatal outcomes in six reference centers in the Northeast of Brazil.

Specific objectives

In pregnant and postpartum women admitted to the four institutions involved with flu-like symptoms or SARS:

1. To describe the biological characteristics (maternal age and pre-pregnancy maternal weight, maternal height, pre-gestational body mass index - BMI and pre-gestational nutritional classification), sociodemographic characteristics (color, number of people living in the household, per capita family income, education, occupation, occupation, marital status, origin and religion), habits (smoking, drinking and use of illicit drugs), obstetric characteristics (number of pregnancies, parity, previous vaginal delivery and previous cesarean, previous abortions, number live children, entry into the study and number of prenatal consultations) and the service of origin (IMIP, HDM, ISEA or MFD);
2. To describe the clinical characteristics (gestational age or postpartum days at the beginning of signs and symptoms, duration of symptoms, isolation, social distance and quarantine before signs and symptoms, need for hospitalization due to infection and / or complications, day of hospitalization due to flu-like syndrome and / or complications, length of hospital stay due to flu-like syndrome and / or complications and the main related signs and symptoms and days of onset - dry or productive cough, runny nose, sore throat, body pain, abdominal pain , chest pain, headache, smell and taste changes, dyspnoea, subfebrile state and fever, diarrhea, asthenia, saturation level, axillary temperature and mild / moderate signs and symptoms);
3. To determine the frequency of COVID-19 infection according to the results of diagnostic tests (rapid test, RT-PCR and serology) applied during hospitalization;
4. To describe the maternal laboratory parameters at the time of the diagnosis of influenza syndrome and the worst laboratory tests (result of RT-PCR for COVID-19, result of viral panel and type of virus, serology for COVID-19 - IgM, IgA and serial IgG, inflammatory cytokines - interleukins - IL-1ra, IL-6, IL-2, IL-5, IL-10, IL-12, IL-13, IL17A, IL-4, IL-1β, IL-9, IL-15, Interferon - IFN-γ, tumor necrosis factor - TNF-α, blood count, coagulogram, urea, creatinine, transaminases - ALT, AST, erythrocyte sedimentation rate - VSH, C reactive protein - CRP), D-dimer, lactic dehydrogenase - LDH, alkaline phosphatase, bilirubins, ferritin, troponin, blood culture, urine culture, blood gas analysis and day of all tests);
5. To describe the radiological findings (chest X-rays, computed tomography), the pulmonal ultrasonography and day of exam alteration and normalization;
6. To describe the therapeutic modalities performed (oxygen therapy - nasal catheter or Venturi with its maximum flows, use of prone in spontaneous ventilation and / or mechanical ventilation, use of mechanical ventilation, use of neuromuscular blocker, use of extracorporeal membrane oxygenation - ECMO, use of: antibiotics, azithromycin, hydroxychloroquine / chloroquine, antiparasitic drugs such as ivermectin, anticoagulant and / or antiretroviral, pulse therapy, convalescent plasma, need for renal replacement therapy, blood products and others, start day and duration of all therapeutic modalities performed);
7. To describe the characteristics of obstetric ultrasound (tachycardia, frequency of diagnosis of fetal growth restriction, fetus small for gestational age - SGA, changes in amniotic fluid and fetal morphological changes) performed during the course of infection and post-infection follow-up;
8. To describe the doppler velocimetric parameters of the uterine and fetal circulation (pulsatility index of the middle uterine arteries, the middle fetal cerebral artery - MCA, the umbilical artery, the venous duct, the frequency of changes in the doppler velocimetry of all the vessels studied and the speed of the systolic peak in MCA) during infection and in the post-infection follow-up;
9. To describe invasive intrauterine diagnostic procedures (amniocentesis), gestational age at which amniocentesis was performed, indications, results of the RT-PCR test for COVID-19, results of the TORCHS survey, results of the karyotype and results of the inflammatory cytokines - interleukins - IL-1ra, IL-6, IL-2, IL-5, IL-10, IL-12, IL-13, IL17A, IL-4, IL-1β, IL-9, IL-15, Interferon - IFN- γ, tumor necrosis factor - TNF-α;
10. To determine comorbidities / complications associated with pregnancy or the puerperium (need for hospitalization due to obstetric causes, length of hospital stay, obesity, multiple pregnancy, hypertensive syndromes, diabetes - clinical or gestational, heart disease, chronic obstructive pulmonary disease, bronchial asthma, cerebrovascular disease, renal failure, immunosuppression, severe acute respiratory syndrome - SARS, premature rupture of membranes, premature labor, placenta praevia, urinary tract infection, pneumonia, sepsis, septic shock, abortion, abruptio placenta, postpartum hemorrhage, infection of surgical site, endometritis, peritonitis, thromboembolic events, need for postpartum hysterectomy, need for other surgeries after delivery and tubal ligation, maternal near miss criteria);
11. To describe the delivery outcomes (type of delivery - vaginal, spontaneous or operative, or cesarean section, indication for cesarean section, indication for labor induction, method of labor induction, duration of induction, gestational age at delivery, use of labor analgesia, type of anesthesia for cesarean section);
12. To describe prenatal interventions (antenatal corticosteroid therapy - number of doses, use of magnesium sulfate and prophylactic antibiotic therapy);
13. To describe the final maternal outcome (discharge of the pregnant woman, discharge of the postpartum woman, death of the pregnant woman and death of the postpartum woman);
14. To describe perinatal and neonatal outcomes (fetal death, perinatal death, birth weight, birth weight adequacy - SGA, AGA, LGA, Apgar scores in the first and fifth minutes, need for neonatal resuscitation, ICU admission, need for assisted mechanical ventilation, oxygen therapy, oxygen therapy modalities, hypothermia, hypoglycemia, polycythemia, anemia, neonatal infection, chorioamnionitis, type of respiratory distress, breastfeeding, neonatal congenital infections (TORCHS), congenital malformation, other neonatal morbidities, neonatal near miss, neonatal death, days of life of neonatal death and length of hospital stay and in neonatal ICU);
15. To determine the procedures in neonatal care in the delivery room (cord clamping - early or opportune, skin-to-skin contact, breastfeeding in the delivery room) and, subsequently, rooming-in or admission to a neonatal ICU / nursing unit;
16. To describe the neonatal laboratory parameters of the suspected diagnosis or confirmation of COVID-19 and the worst test results (days of life of the newborn's suspected diagnosis, result of rapid neonate test, RT-PCR for COVID-19 in nasopharyngeal swab , result of viral panel and virus type, serology for COVID-19 - IgM, IgA and IgG serial, inflammatory cytokines - interleukins - IL-1ra, IL-6, IL-2, IL-5, IL-10, IL -12, IL-13, IL17A, IL-4, IL-1β, IL-9, IL-15, Interferon - IFN-γ, tumor necrosis factor - TNF-α, blood count, coagulogram, urea, creatinine, transaminases - ALT, AST, erythrocyte sedimentation rate - VSH, C-reactive protein - CRP), D-dimer, lactic dehydrogenase - LDH, alkaline phosphatase, bilirubins, ferritin, troponin, blood culture, urine culture, blood gas analysis and day of all tests);
17. To describe the laboratory parameters in the placenta (result of RT-PCR / viral panel by swab and anatomopathological study) and in cord blood (RT-PCR);
18. To determine the frequency of vertical transmission and the factors associated with a higher risk of its occurrence (gestational age at infection, severity of infection, laboratory markers, type of delivery, labor, cord clamping practice, placental findings, maternal interleukins);
19. To describe the laboratory parameters in breast milk (result of RT-PCR / viral panel);
20. To describe the neonatal imaging exams (chest X-rays, computed tomography and day of exam changes and normalization);
21. To determine the association of biological, sociodemographic, obstetric variables, habits, clinical, maternal laboratory parameters in the diagnosis and the worst result, radiological findings, therapeutic modalities, ultrasound and doppler velocimetric characteristics, invasive procedures, comorbidities / complications and characteristics of childbirth with adverse maternal outcome (maternal near miss and maternal death).
22. To determine the association of biological, sociodemographic, obstetric variables, habits, clinical, maternal laboratory parameters in the diagnosis and the worst result, radiological findings, therapeutic modalities, ultrasound and doppler velocimetric characteristics, invasive procedures, comorbidities / complications, delivery results, prenatal interventions, final pregnancy outcome, delivery room procedures, neonatal care and neonatal laboratory parameters, placenta, amniotic fluid and breast milk with adverse perinatal / neonatal outcome (neonatal near miss and fetal / neonatal death);
23. To analyze maternal and perinatal mortality according to gestational age at the onset of symptoms (Kaplan-Meier survival curve);
24. To compare data from two states in Northeast Brazil with official general data in the country according to the Ministry of Health for the pregnancy-puerperal cycle.
25. In a subset of women routinely assessed on admission through the rapid test (ISEA and Unimed-João Pessoa), to determine the frequency of positive rapid test, positive RT-PCR, associated symptoms, asymptomatic carriers and to compare maternal and perinatal outcomes according to test results.
26. To carry out long-term monitoring of women and babies included in the cohort in 2020, to detect recurrence of symptoms, frequency of reinfection, evolution of laboratory parameters (repetition of RT-PCR and serology) and monitoring of growth and development in the cohort of children aged six months, 12 and 24 months.

Methods: A prospective and retrospective cohort study will be conducted including pregnant and postpartum women with clinical or laboratorial diagnosis of COVID-19, admitted in six healthcare centers in the Northeast of Brazil. All pregnant and postpartum women with clinical and/or diagnosis of COVID-19, attended in prenatal care, in emergency (maternity triage), high-risk pregnancy ward, obstetric intensive care unit and rooming-in ward will be included. The data will be collected in specific forms. The exams will be carried out by trained professionals within each institution. A database will be created on the RedCap platform. For the association of dependent variables (maternal mortality / near miss and unfavorable perinatal outcomes) with independent variables (biological, sociodemographic characteristics, history, clinical characteristics, ultrasound modifications, doppler velocimetric and laboratory tests, chi-square tests will be used and Fisher's exact, when pertinent, with a significance level of 5%. The relative risk and its 95% confidence interval will also be calculated to determine the strength of association between the variables. outcomes, Student t or Mann-Whitney tests will be adopted. A multivariate analysis will be performed to determine the variables that will actually remain associated, in addition, a Kaplan-Meier survival curve will be constructed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or puerperal women;
* Diagnosis of flu syndrome on admission;
* Testing for COVID-19 performed.

Exclusion Criteria:

* Clinical impossibility of signing the Informed Consent Form (ICF), either by the patient or guardian (in the prospective arm);
* Incomplete or not located medical records (retrospective arm).

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant and postpartum women admitted with flu syndrome in six reference centers in the Northeast of Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Near miss maternal: | 42 days
  Refers to a woman who almost died, but survived a serious complication that occurred during pregnancy, childbirth or within 42 days after termination of the pregnancy, depending on the presence of at least one of the criteria adopted by the World Health Organization ( WHO). Variable, categorical and dichotomous yes / no type.
Maternal death | 42 days
  It is the death of a woman during pregnancy or within 42 days after the end of the pregnancy or due to measures taken in relation to the pregnancy, but not due to accidental or incidental causes. Variable, categorical and dichotomous yes / no type.
Near miss neonate | 7 days
  It refers to the newborn classified with severe morbidity by pragmatic criteria (Apgar <7 in the 5th minute, birth weight <1,750 grams or gestational age <33 weeks) or conduct (parenteral antibiotic therapy - up to 7 days and before the 28th day of life, nasal CPAP, intubation, up to 7 days and before the 28th day of life, phototherapy within 24 hours of life, cardiopulmonary resuscitation, use of vasoactive drugs, use of anticonvulsants, use of blood products, use of corticosteroids to treat refractory hypoglycemia and surgery) but who survived the 27th day of life, included. Yes / no categorical and dichotomous variable.
Neonatal death | 27 days
  Death occurred in the first 27 days, included, after delivery. Yes / no categorical and dichotomous variable.
Early neonatal death | 7 days
  Death occurred in the first 7 days of life. Yes / no dichotomous categorical variable
Fetal death | 1 hour
  Intrauterine death, corresponding to the birth of a fetus without signs of life, weighing 500 grams or more. Dichotomous categorical variable of the yes / no type.
Perinatal death | 7 days
  Corresponds to cases of fetal death added to those of early neonatal death. Dichotomous categorical variable of the yes / no type.

SECONDARY OUTCOMES:
Maternal age | 1 hour
  Calculated based on the date of birth recorded in the medical record, hospital identification data, or according to the patient's information, in full years. Numerical and discrete variable.
Maternal pre-pregnancy weight | 1 hour
  maternal weight before pregnancy, in kilogram (kg), according to information collected from the patient and / or made available on the prenatal card or medical record. Numeric and continuous variable.
Maternal height | 1 hour
  expressed, in meters, according to information collected from the patient and / or made available on the prenatal card or medical record. Numeric and continuous variable.
Pre-gestational nutritional classification | 1 hour
  classified according to pre-gestational BMI: low weight grade III (≤ 16.00), low weight grade II (≥ 16.00 to <16.99), low weight grade I (≥ 17 , 00 to <18.49), ideal weight (≥ 18.50 to <24.99), overweight (≥ 25.00 to <29.99), grade I obesity (≥ 30.00 to <34.99) , grade II obesity (≥35.00 to <39.99) and grade III obesity (≥ 40.00).
Pre-gestational body mass index (BMI) | 1 hour
  expressed in Kg / m2, calculated by weight (kg) divided by height (m) squared. Numeric and continuous variable.
Maternal color | 1 hour
  according to the patient's self-declaration and collected according to information and / or recorded in the medical record or prenatal card in black, white, brown, yellow and indigenous.
Number of people living in the household | 1 hour
  defined as the number of people, regardless of age, living in the same household, collected according to the patient's information. Numerical and discrete variable.
Family income per capita | 1 hour
  collected according to the patient's information as the sum of the monthly income of all members living in the household, including benefits from social programs and informal income. Categorized in: up to 1 minimum wage; 1 to 2 minimum wages; 3 to 5 minimum wages; more than 5 minimum wages. Numerical and discrete variable.
Maternal education | 1 hour
  as informed by the patient, recorded in medical records or prenatal card and categorized as illiterate (zero), elementary school (one to nine years), high school (10 to 12 years) and higher education (> 12 years) ). Numerical and discrete variable.
Maternal occupation | 1 hour
  as declared by the patient and noted on the medical record or prenatal card, later categorized as: health, education, general services, home, domestic, student, merchant or commerce, security, self-employed, economy, tourism, music, nutrition, computers, journalism, engineering and others.
Maternal occupation with financial income | 1 hour
  as declared by the patient, as being a formal job or not, which presents any monthly financial income. Yes / no categorical and dichotomous variable.
Maternal marital status | 1 hour
  declared by the patient and recorded in medical records or prenatal card in: single, married, stable, separated and widowed.
Maternal origin | 1 hour
  as informed by the patient and recorded in medical records, related to the city where she lives, defined as Recife, metropolitan region (Jaboatão dos Guararapes, Olinda, Paulista, Moreno, Igarassu, Abreu e Lima, Camaragibe, Cabo de Santo Agostinho, São Lourenço da Mata, Araçoiaba, Itamaracá Island, Ipojuca and Itapissuma), interior and other states.
Maternal religion | 1 hour
  according to the belief declared by the patient and categorized into: atheist, catholic, evangelical, spiritist, Anglican charismatic and others.
Maternal smoking | 1 hour
  smoking, regardless of quantity, during pregnancy, as stated by the patient. Yes / no categorical and dichotomous variable.
Maternal alcoholism | 1 hour
  habit of drinking alcoholic beverages, regardless of quantity, during pregnancy, as stated by the patient. Yes / no categorical and dichotomous variable.
Maternal use of illicit drugs | 1 hour
  use of non-legal drugs, such as marijuana, cocaine, crack and the like, regardless of the amount, during pregnancy, as stated by the patient. Yes / no categorical and dichotomous variable.
Number of pregnancies | 1 hour
  number of previous pregnancies, including the current one, regardless of the gestational outcome (abortion, delivery, number of fetuses, ectopic pregnancy or fetal death), as reported by the patient and noted in the medical record or prenatal card. Numerical and discrete variable.
Parity | 1 hour
  number of previous deliveries with fetuses over 500g and / or gestational age greater than 22 weeks, regardless of multiple gestation, perinatal death or delivery, as reported by the patient and noted in the medical record or prenatal card. Numerical and discrete variable.
Number of previous cesarean sections | 1 hour
  number of previous deliveries with fetuses over 500g and / or gestational age greater than the 22nd week, by cesarean section, as informed by the patient and noted in the medical record or prenatal card. Numerical and discrete variable.
Number of previous vaginal births | 1 hour
  number of previous births with fetuses above 500g and / or gestational age greater than 22 weeks, vaginally, regardless of whether instrumental, as informed by the patient and noted in the medical record or prenatal card. Numerical and discrete variable.
Number of previous abortions | 1 hour
  number of interruptions of pregnancy with fetuses below 500g and / or gestational age below 22 weeks, regardless of being spontaneous, as informed by the patient and noted in the medical record or prenatal card. Numerical and discrete variable.
Number of children alive | 1 hour
  number of children who remain alive, regardless of the cause of death, as informed by the patient and noted in medical records or prenatal card. Numerical and discrete variable.
Number of prenatal consultations | 1 hour
  as informed by the patient or noted on the prenatal card and medical record, the number of consultations performed during prenatal care. Numerical and discrete variable.
Gestational age of the onset of flu-like signs and symptoms | 1 hour
  gestational age, in weeks, calculated by the day of the last menstruation and confirmed by the first ultrasound scan of the onset of flu-like signs and symptoms. Numerical and discrete variable.
Number of puerperium days of onset of flu-like signs and symptoms | 14 days
  number of days after birth of the onset of flu-like signs and symptoms. Numerical and discrete variable.
Duration of maternal symptoms | 1 hour
  number of days the patient had signs and symptoms of flu-like syndrome and its complications. Numerical and discrete variable.
Social isolation during the signs and symptoms of flu-like syndrome | 14 days
  when the patient declared that at the beginning of the signs and symptoms she was separated / isolated at home without any contact with healthy people, including not even going out for essential purchases, for a period of 14 days. Yes / No categorical and dichotomous variable.
Social distance before the signs and symptoms of flu-like syndrome | 1 hour
  it is a measure of community restraint, adopted in some cases, to prevent the spread of a certain contagious disease. Considered when the patient declared that she was at home, leaving only what was necessary for essential purchases, before the onset of signs and symptoms. Yes / No categorical and dichotomous variable.
Quarantine | 14 days
  when the patient declared that she had contact with people infected with COVID-19 and / or traveled to places considered to be the epicenter of the disease, but even asymptomatic, she stayed home without contact with other people, including not even going out for essential purchases, for a period of seven to 14 days. Yes / No categorical and dichotomous variable.
Need for hospitalization due to flu-like syndrome and/or complications | 1 hour
  when there is a need for hospitalization due to flu-like syndrome and / or its complications, excluding hospitalizations due to obstetric complications and includes all participants, especially pregnant women monitored during prenatal care. Yes / No categorical and dichotomous variable.
Day of hospitalization due to flu syndrome and/or complications | 1 hour
  day of hospitalization due to flu syndrome and / or complications. Numerical and discrete variable.
Length of hospital stay due to flu-like syndrome and/or complications | 14 days
  length of stay, in days, as described in the medical record. Numerical and discrete variable.
Maternal signs and symptoms of flu-like syndrome at diagnosis, at 6 months, 12 months and 24 months | 24 months
  As reported by the patient (dry cough, day of onset of dry cough, productive cough, day of onset of productive cough, coryza, day of onset of runny nose, body pain, day of onset of body pain, abdominal pain, day of onset of abdominal pain, chest pain, day of onset of chest pain, headache, day of onset of headache, dyspnoea, day of onset of dyspnoea, subfebrile state, day of onset of subfebrile state, fever, day of onset of fever, diarrhea , day of onset of diarrhea, sore throat, day of onset of sore throat, taste change, day of onset of taste change, smell change, day of onset of smell change, asthenia, day of onset of asthenia , axillary temperature, oxygen saturation).
Result of polymerase chain reaction - real time (RT-PCR) for maternal COVID19 in diagnosis, at 6 months, 12 months and 24 months | 24 months
  result of RT-PCR in the diagnosis of COVID-19, by means of blood or nasopharyngeal secretion, according to the usual technique, being categorized as positive, negative and indeterminate.
Result of polymerase chain reaction - real time (RT-PCR) for the differential diagnosis of maternal respiratory syndrome (viral panel) | 10 days
  result of RT-PCR in the differential diagnosis of respiratory syndrome, through blood or nasopharyngeal secretion, according to the technique and kit used, being categorized as positive (any virus found), negative and indeterminate.
Maternal viral panel in the diagnosis, at 6 months, 12 months and 24 months | 24 months
  result of the RT-PCR of the viral panel in the differential diagnosis of flu syndrome, through blood or nasopharyngeal secretion, according to the technique and kit used, categorized according to the virus found.
Rapid test for maternal COVID-19 at diagnosis, at 6 months, 12 months and 24 months | 24 months
  result in the diagnosis of COVID-19, by means of blood, according to the usual technique, being categorized as positive, negative and indeterminate.
Serial maternal IgM COVID-19 | 6 months, 12 months and 24 months
  result of IgM COVID-19 serology, through blood, according to the Enzyme-Linked Immunosorbent Assay (ELISA) technique or immunochromatography or chemiluminescent immunoassay, being categorized as positive, negative and indeterminate, according to the reference values of each serological kit, performed after the 5th day of signs and symptoms. Numeric and continuous variable.
Serial maternal IgA COVID-19 | 6 months, 12 months and 24 months
  result of IgA COVID-19 serology, through blood, according to the ELISA technique, being categorized as positive, negative and indeterminate, according to the reference values of each serological kit, performed after 5th day of signs and symptoms. Numeric and continuous variable.
Serial maternal IgG COVID-19 | 6 months, 12 months and 24 months
  result of IgG COVID-19 serology, by means of blood, according to the ELISA technique, being categorized as positive, negative and indeterminate, according to the reference values of each serological kit, performed after 14th day of signs and symptoms. Numeric and continuous variable.
Serial maternal serology day | 6 months, 12 months and 24 months
  rom the first exam (day zero). Describe the subsequent days. Numerical and discrete variable.
Maternal reinfection | 14 days
  after diagnostic confirmation of COVID-19 and 14 days after the cure criteria, the RT-PCR test returns positive. Yes / No categorical and dichotomous variable.
Cytokines in maternal diagnosis | 14 days
  substances capable of modulating the cellular response of several cells, such as interleukins - IL-1ra, IL-6, IL-2, IL-5, IL-10, IL-12, IL-13, IL17A, IL-4, IL-1β, IL-9, IL-15, Interferon - IFN-γ and Tumor necrosis factor - TNF-α, in maternal blood, in pg / ml, from the beginning of the flu syndrome or COVID- 19 and in the period of the syndrome. Numeric and continuous variable (for each cytokine).
Day of the first cytokine dosage from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the first cytokine dosage from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
Day of the first blood count from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the first blood count from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
Hemoglobin of maternal diagnosis | 14 days
  value of the first hemoglobin measured in maternal blood, in g / dL, from the flu syndrome and in the period of the syndrome, being normal ≥ 11.0g / dL and ≤ 16.0g / dL. Numeric and continuous variable.
Leukocytes from maternal diagnosis | 14 days
  value of the first leukocyte measured in maternal blood, / mm3, from the flu syndrome and in the period of the syndrome, being normal ≥ 4,000 / mm3 and ≤ 11,000 / mm3. Numerical and discrete variable.
Deviation to the left of the maternal diagnosis | 14 days
  when the rod / segment ratio is greater than 1/16 and / or the presence of young cells (promyelocytes, myelocytes, metamyelocytes) occurs, starting with the flu syndrome and in the period of the syndrome. Yes / No categorical and dichotomous variable.
Platelets of maternal diagnosis | 14 days
  value of the first platelet measured in maternal blood, / mm3, from the flu syndrome and in the period of the syndrome, being normal ≥ 150,000 / mm3 and ≤ 400,000 / mm3. Numerical and discrete variable.
Typical lymphocytes of maternal diagnosis | 14 days
  value of the first typical lymphocyte measured in maternal blood, / mm3, from the flu syndrome and in the period of the syndrome, being normal ≥ 1,050 / mm3 and ≤ 3,850 / mm3. Numerical and discrete variable.
Atypical lymphocytes of maternal diagnosis | 14 days
  value of the first atypical lymphocyte measured in maternal blood, / mm3, from the flu syndrome and in the period of the syndrome, being normal ≥ 0 / mm3 and ≤ 220 / mm3. Numerical and discrete variable.
Day of the first coagulogram from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the first coagulogram from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
Maternal diagnosis bleeding time (TB) | 14 days
  value of the first TB measured in maternal blood, in seconds (s), from the flu syndrome and the period of the syndrome, being normal from 60s to 180s. Numerical and discrete variable.
Maternal diagnosis clotting time (CT) | 14 days
  value of the first CT measured in maternal blood, in seconds (s), from the flu syndrome and the period of the syndrome. Numerical and discrete variable.
Maternal prothrombin time of diagnosis (TD) | 14 days
  value of the first TD measured in maternal blood, in seconds (s), from the flu syndrome and in the period of the syndrome, with a value of up to 11.3s being normal. Numerical and discrete variable.
Maternal active partial thromboplastin time of diagnosis (APTT) | 14 days
  value of the first APTT measured in maternal blood, in seconds (s), from the flu syndrome and the period of the syndrome, with a value of up to 30.5s being normal.
International normalized ratio (INR) | 14 days
  value of the first INR measured in maternal blood, from the flu syndrome and the period of the syndrome, being normal between 2 and 3. Numerical and discrete variable.
Day of the first urea from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the first urea from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
Urea from maternal diagnosis | 14 days
  value of the first urea measured in maternal blood, in mg / dL, from the flu syndrome and in the period of the syndrome, being normal ≥ 19.2mg / dL and ≤ 49.2mg / dL. Numerical and discrete variable.
Day of the first creatinine from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the first creatinine from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
Creatinine of maternal diagnosis | 14 days
  value of the first creatinine measured in maternal blood, in mg / dL, from the flu syndrome and in the period of the syndrome, being normal ≥ 0.5mg / dL and ≤ 1.1mg / dl. Numerical and discrete variable.
Transaminases in maternal diagnosis | 14 days
  defined as aspartate aminotransferase (AST) or glutamic-oxalacetic transaminase (TGO) and alanine aminotransferase (ALT) or glutamic-pyruvic transaminase (TGP), from the beginning of the flu syndrome or COVID-19 on syndrome period.
Day of the first erythrocyte sedimentation rate (VSH) of maternal diagnosis from the beginning of the flu syndrome or COVID-19: | 14 days
  day of the first VSH from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
VSH of maternal diagnosis | 14 days
  value of the first VSH measured in maternal blood, in mm / h, from the flu syndrome and in the period of the syndrome, being normal <20mm / h. Numerical and discrete variable.
Day of the first C-reactive protein (CRP) from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the first CRP from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
CRP of maternal diagnosis | 14 days
  value of the first CRP measured in maternal blood, in mg / L, from the flu syndrome and in the period of the syndrome, being normal <5mg / L. Numerical and discrete variable.
Day of the first D-dimer from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the first D-dimer from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
D-dimer of maternal diagnosis | 14 days
  value of the first D-dimer dosed in maternal blood, in mg / dL, from the flu syndrome and the period of the syndrome. Numerical and discrete variable.
Day of the first lactic dehydrogenase (DHL) from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the first DHL from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
DHL of maternal diagnosis | 14 days
  value of the first DHL measured in maternal blood, in mg / dL, from the flu syndrome and the period of the syndrome, being normal ≥ 125U / L and ≤ 243U / L. Numerical and discrete variable.
Day of the first alkaline phosphatase from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the first alkaline phosphatase from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
Alkaline phosphatase in maternal diagnosis | 14 days
  value of the first alkaline phosphatase measured in maternal blood, in U / L, from the flu syndrome and in the period of the syndrome, being normal ≥ 46U / L and ≤ 116U / L. Numerical and discrete variable.
Day of the first troponin from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the first troponin from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
Troponin in maternal diagnosis | 14 days
  value of the first troponin measured in maternal blood, in ng / mL, from the flu syndrome and in the period of the syndrome, being normal <0.4 ng / mL. Numerical and discrete variable.
Day of the first ferritin from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the first ferritin from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
Ferritin in maternal diagnosis | 14 days
  alue of the first ferritin measured in maternal blood, in ng / mL, from the flu syndrome and the period of the syndrome. Numerical and discrete variable.
Bilirubins in maternal diagnosis | 14 days
  defined as total (BT), direct (BD) and indirect (BI) bilirubins from the beginning of the flu syndrome or COVID-19 and in the period of the syndrome.
Day of the first blood culture from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the first blood culture from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
Blood culture of maternal diagnosis | 14 days
  result of the first blood culture from the flu syndrome and in the period of the syndrome, categorized as negative and positive (growth of the microorganism). Categorical and dichotomous variable.
Blood culture microorganism in maternal diagnosis | 14 days
  name of the microorganism, which grew on examination, from the flu syndrome and the period of the syndrome, according to its taxonomic classification.
Day of the first uroculture from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the first uroculture from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
Uroculture of maternal diagnosis | 14 days
  result of the first uroculture from the flu syndrome and in the period of the syndrome, categorized as negative and positive (growth of the microorganism). Categorical and dichotomous variable.
Uroculture microorganism in maternal diagnosis | 14 days
  name of the microorganism, which grew on examination, from the flu syndrome and the period of the syndrome, according to its taxonomic classification.
IgM COVID-19 worst maternal result | 5 days
  worst result of IgM COVID-19 serology, through blood, according to the Enzyme-Linked Immunosorbent Assay (ELISA) technique or immunochromatography or chemiluminescent immunoassay, being categorized as positive, negative and indeterminate, of according to the reference values of each serological kit, performed after the 5th day of signs and symptoms. Numeric and continuous variable.
IgA COVID-19 worst maternal result | 5 days
  Result of the worst result of IgA COVID-19 serology, through blood, according to the ELISA technique, being categorized as positive, negative and indeterminate, according to the reference values of each serological kit , performed after the 5th day of signs and symptoms. Numeric and continuous variable.
Maternal IgG COVID-19 - worst serial result | 14 days
  worst result of IgG COVID-19 serology, performed using blood, according to the ELISA technique, being categorized as positive, negative and indeterminate, according to the reference values of each kit serological test, performed after the 14th day of signs and symptoms. Numeric and continuous variable.
Cytokines worst maternal outcome | 14 days
  substances capable of modulating the cellular response of several cells, such as interleukins - IL-1ra, IL-6, IL-2, IL-5, IL-10, IL-12, IL-13, IL17A , IL-4, IL-1β, IL-9, IL-15, Interferon - IFN-γ and Tumor necrosis factor - TNF-α, in maternal blood, in pg / ml, being the worst maternal result, from the beginning of the flu syndrome or COVID-19 and in the period of the syndrome. Numeric and continuous variable (for each cytokine).
Day of the worst urea result from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the performance of the worst urea result from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
Urea worst maternal result | 14 days
  value of the worst result of urea measured in maternal blood, in mg / dL, from the flu syndrome and in the period of the syndrome being normal ≥ 19.2mg / dL and ≤ 49.2mg / dL. Numerical and discrete variable.
Day of the worst creatinine result from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the worst creatinine result from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
Creatinine worst maternal result | 14 days
  value of the worst result of creatinine measured in maternal blood, in mg / dL, from the flu syndrome and in the period of the syndrome, being normal ≥ 0.5mg / dL and ≤ 1.1mg / dl. Numeric and discrete variable.
Transaminases worst maternal outcome | 14 days
  defined as the worst outcome of aspartate aminotransferase (AST) or glutamic-oxalacetic transaminase (TGO) and alanine aminotransferase (ALT) or glutamic-pyruvic transaminase (TGP) from the onset of the flu syndrome or COVID- 19 and in the period of the syndrome.
Day of the worst result of the erythrocyte sedimentation rate of maternal diagnosis (VSH) from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the worst VSH result from the flu syndrome and the period of the syndrome. Numerical and discrete variable.
VSH worst maternal result | 14 days
  value of the worst result of VSH measured in maternal blood, in mm / h, from the flu syndrome and in the period of the syndrome, being normal <20mm / h. Numerical and discrete variable.
Day of the worst C-reactive protein (CRP) result from the onset of the flu syndrome or COVID-19 | 14 days
  day of the worst CRP result from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
CRP worst maternal result | 14 days
  value of the worst CRP result measured in maternal blood, in mg / L, from the flu syndrome and in the period of the syndrome, being normal <5mg / L. Numerical and discrete variable.
Day of the worst D-dimer result from the onset of the flu syndrome or COVID-19 | 14 days
  day of the worst D-dimer result from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
D-dimer worst maternal result | 14 days
  value of the worst D-dimer result measured in maternal blood, in mg / dL, from the flu syndrome and the period of the syndrome. Numerical and discrete variable.
Day of the worst result of lactic dehydrogenase (DHL) from the beginning of the flu syndrome or COVID-19 | 14 days
  day of the worst DHL result from the flu syndrome and in the period of the syndrome. Numerical and discrete variable.
DHL worst maternal result | 14 days
  value of the worst DHL result measured in maternal blood, in mg / dL, from the flu syndrome and the period of the syndrome, being normal ≥ 125U / L and ≤ 243U / L. Numerical and discrete variable.
Alkaline phosphatase worst maternal result | 14 days
  value of the worst result of alkaline phosphatase measured in maternal blood, in U / L, from the flu syndrome and in the period of the syndrome, being normal ≥ 46U / L and ≤ 116U / L. Numerical and discrete variable.
Troponin worst maternal result | 14 days
  value of the worst result of troponin dosed in maternal blood, in ng / mL, from the flu syndrome and in the period of the syndrome, being normal <0.4 ng / mL. Numerical and discrete variable.
Ferritin worst maternal result | 14 days
  value of the worst result of ferritin measured in maternal blood, in ng / mL, from the flu syndrome and the period of the syndrome. Numerical and discrete variable.
Bilirubins worst maternal result | 14 days
  defined as the worst result of total (BT), direct (BD) and indirect (BI) bilirubins from the beginning of the flu syndrome or COVID-19 and in the period of the syndrome.
Blood culture worst maternal result | 14 days
  result of the worst blood culture from the flu syndrome and in the period of the syndrome, categorized as negative and positive (growth of the microorganism). Categorical and dichotomous variable.
Blood culture microorganism worst maternal result | 14 days
  name of the microorganism, which grew on the exam, in the worst maternal result, from the flu syndrome and the period of the syndrome, according to its taxonomic classification.
Uroculture worse maternal result | 14 days
  result of the worst uroculture from the flu syndrome and in the period of the syndrome, categorized as negative and positive (growth of the microorganism). Categorical and dichotomous variable.
Uroculture microorganism worst maternal result | 14 days
  name of the microorganism, which grew in the exam, in the worst maternal result, from the flu syndrome and the period of the syndrome, according to its taxonomic classification.
Presence of changes in maternal chest radiography | 14 days
  presence of any radiological changes, described in a medical report. Yes / No categorical and dichotomous variable.
Result of maternal chest radiography | 14 days
  description of any radiological alterations, described in a medical report.
Presence of changes in the mother's chest tomography | 14 days
  presence of any changes in the tomography described in a medical report. Yes / No categorical and dichotomous variable.
Day of normalization of the alteration of the tomography of the maternal chest | 14 days
  day of the normalization of any alteration of the tomography, described in a medical report, as of the appearance. Numerical and discrete variable.
Result of maternal chest tomography | 14 days
  description of any alteration of the tomography described in a medical report.
Use of maternal nasal catheter | 1 month
  need for maternal nasal catheter to maintain normal oxygen saturation. Yes / No categorical and dichotomous variable.
Use of maternal Venturi Mask | 1 month
  need for Venturi mask to maintain normal oxygen saturation. Yes / No categorical and dichotomous variable.
Prone maternal position on spontaneous ventilation | 1 month
  when the patient was placed in prone position on spontaneous ventilation, face down, which was used to improve oxygenation. Yes / No categorical and dichotomous variable.
Use of therapeutic antibiotics | 14 days
  need for antibiotic therapy to treat associated bacterial infection. Yes / No categorical and dichotomous variable.
Use of azithromycin | 14 days
  need for azithromycin as a complementary treatment for COVID-19. Yes / No categorical and dichotomous variable.
Use of maternal hydroxychloroquine/chloroquine | 14 days
  need for hydroxychloroquine / chloroquine as a complementary treatment for COVID-19. Yes / No categorical and dichotomous variable.
Use of antiparasitic drugs | 14 days
  need for antiparasitic drugs as a complementary treatment for COVID-19. Yes / No categorical and dichotomous variable.
Use of anticoagulant | 14 days
  need for anticoagulant as a complementary treatment for COVID-19. Yes / No categorical and dichotomous variable.
Use of antiretroviral | 14 days
  need for antiretroviral as a complementary treatment for COVID-19. Yes / No categorical and dichotomous variable.
Use of pulse therapy | 14 days
  need for corticosteroid pulse therapy as a complementary treatment for COVID-19. Yes / No categorical and dichotomous variable.
Use of convalescent plasma | 14 days
  need for patient-cured plasma from COVID-19 (convalescent) as a complementary treatment to COVID-19. Yes / No categorical and dichotomous variable.
Assisted Mechanical Ventilation (AMV) | 1 month
  need for AMV as a complementary treatment to COVID-19. Yes / No categorical and dichotomous variable.
Use of neuromuscular blocker | 14 days
  need for medication for neuromuscular block, such as pancuronium, as assessed by the attending physician and described in the medical record. Yes / No categorical and dichotomous variable.
Use of Extracorporeal Circulation (ECMO) | 1 month
  need to use ECMO to better oxygenate the lungs and heart. Yes / No categorical and dichotomous variable.
Renal replacement therapy (dialysis) | 1 month
  need for dialysis (peritoneal or hemodialysis) as a complementary treatment for COVID-19. Yes / No categorical and dichotomous variable.
Blood products | 1 month
  need for blood products as a complementary treatment to COVID-19. Yes / No categorical and dichotomous variable.
Other therapeutic modalities | 1 month
  need for other complementary treatments of COVID-19. Yes / No categorical and dichotomous variable.
Amniotic fluid in the last ultrasound examination | 14 days
  defined by the amniotic fluid index (ILA) or the largest pocket, according to the experience of the ultrasonographer. The ILA will be measured in cm, being defined as the sum of the largest pockets of amniotic fluid in the four quadrants of the maternal abdomen. It will be categorized into: normal (between 8.0 and 18.0cm), decreased (between 7.9 and 5.0cm), moderate oligohydramnios (between 4.9 and 3.0cm), severe oligohydramnios (<3 , 0cm), increased (between 18.1 and 24cm) and polyhydramnios (ILA> 24cm) (81.82). The largest pocket will also be measured in cm, being defined as the measure of the largest pocket of amniotic fluid in the four quadrants of the maternal abdomen. It will be categorized into: normal (between 3.0 and 8.0cm), decreased (between 2.9 and 2.0cm), moderate oligoamine (between 1.9 and 1.0cm), severe oligoamine (<1.0cm), increased (ILA between 8.1 and 12.0cm) and polyhydramnios (ILA> 12.0cm).
Fetal growth restriction | 14 days
  defined by the Delphi procedure 2016 . Yes / No categorical and dichotomous variable.
Small fetus for gestational age (SGA) | 14 days
  defined when the estimated fetal weight is <10pct for gestational age and does not meet the criteria for IUGR. Yes / No categorical and dichotomous variable.
Presence of fetal morphological changes | 1 month
  presence of any abnormalities in fetal formation, major defects, or presence of minor changes diagnosed by ultrasound. Yes / No categorical and dichotomous variable.
Fetal morphological changes | 1 month
  description of any abnormalities in fetal formation, major defects, or presence of minor changes diagnosed by ultrasound.
Frequency of fetal tachycardia (FFT) | 1 month
  increased FFT diagnosed by ultrasound or Doppler sonar, with sinus rhythm, when greater than 160bpm. Yes / No categorical and dichotomous variable.
Doppler velocimetry parameters in the last ultrasound examination | 1 month
  from the pulsatility index (PI), which is automatically calculated by the ultrasound device, using the formula: systolic peak minus the diastolic peak divided by the average speed.
Gestational age of amniocentesis | 1 month
  gestational age, in weeks, calculated by the day of the last menstruation and confirmed by the first ultrasound of amniocentesis. Numerical and discrete variable.
Amniocentesis indications | 1 month
  indication for amniocentesis, due to COVID-19 or another cause.
Result of amniocentesis for COVID19 | 1 month
  result of RT-PCR for COVID-19, in amniotic fluid, according to the usual technique, being categorized as positive, negative and indeterminate.
Amniocentesis cytokines | 1 month
  substances capable of modulating the cellular response of several cells, such as interleukins IL-1ra, IL-6, IL-2, IL-5, IL-10, IL-12, IL-13, IL17A, IL -4, IL-1β, IL-9, IL-15, Interferon - IFN-γ and Tumor necrosis factor - TNF-α, in amniotic fluid, in pg / ml, from the beginning of the flu syndrome or COVID-19 , and in the period of the syndrome. Numeric and continuous variable (for each cytokine).
Need for hospitalization due to obstetric causes | 1 month
  need for hospitalization due to some comorbidity or obstetric complications. Yes / No categorical and dichotomous variable.
Maternal hospital stay | 1 month
  total hospital stay for any comorbidity or obstetric complications. Numerical and discrete variable.
Obesity | 1 month
  calculated based on the last BMI (weight [kg] / height [m] 2), by gestational age, using the curve by Atalah et al. Yes / No categorical and dichotomous variable.
Chronic arterial hypertension (CAH) | 1 month
  defined as blood pressure (BP) greater than or equal to 140 / 90mmHg, diagnosed before pregnancy, or before the 20th week of pregnancy . Yes / No categorical and dichotomous variable.
Superimposed preeclampsia | 1 month
  defined as CAH associated with signs of severity . Yes / No categorical and dichotomous variable.
Gestational hypertension | 1 month
  defined as BP greater than or equal to 140 / 90mmHg, diagnosed above the 20th week of pregnancy, with no signs of severity or proteinuria . Yes / No categorical and dichotomous variable.
Pre-eclampsia | 1 month
  defined as BP greater than or equal to 140 / 90mmHg, above the 20th week of pregnancy, associated with proteinuria (greater than 300mg / dl in 24-hour urine or tape, or protein / creatinine ratio greater than 0.3 ), or target organ dysfunction, which can be categorized as severe and non-severe . Yes / No categorical and dichotomous variable.
Eclampsia | 1 month
  defined as BP greater than or equal to 140 / 90mmHg above the 20th week of gestation, in the presence of proteinuria (greater than 300mg / dl in 24-hour urine or tape, or protein / creatinine ratio greater than 0.3), associated with seizures. Yes / No categorical and dichotomous variable.
HELLP syndrome | 1 month
  defined by the presence of hemolysis, elevated liver enzymes, decreased platelets (below 100,000 / L), elevated TGO / TGP (above 70UI / L) . Yes / No categorical and dichotomous variable.
Clinical diabetes | 1 month
  defined by the presence of one of the criteria: HbA1C ≥ 6.5% or fasting blood glucose ≥ 126mg / dl - the test should be repeated - or random blood glucose> 200mg / dl, associated with symptoms of diabetes , depending on diagnosis declared by the patient and recorded in medical records. Yes / No categorical and dichotomous variable.
Gestational diabetes | 1 month
  defined by the presence of at least one of the criteria after an oral glucose tolerance test (TOTG) performed between the 24th and 28th weeks of gestation: fasting glucose ≥ 92mg / dl, or ≥ 180mg / dl (after one hour), or ≥ 153mg / dl (after two hours) , according to the diagnosis declared by the patient and recorded in medical records. Yes / No categorical and dichotomous variable.
Premature rupture of membranes | 1 month
  spontaneous rupture of the membranes, diagnosed by anamnesis and clinical examination of the pregnant woman, before the start of labor. Yes / No categorical and dichotomous variable.
Premature labor | 1 month
  defined as the spontaneous triggering of labor before term (<37 weeks), when there were above three contractions in 30 minutes and cervical alteration, according to clinical and obstetric evaluation. Yes / No categorical and dichotomous variable.
Placenta previa | 1 month
  define when the placental insertion is low, close to the cervix, regardless of its classification (total, partial and marginal), according to ultrasound report. Yes / No categorical and dichotomous variable.
Abortion | 1 month
  termination of pregnancy before the 22nd week and / or below 500 g, gestational age preferable, provided it is reliable, regardless of whether it is spontaneous or provoked. Yes / No categorical and dichotomous variable.
Normally inserted placental abruption | 1 month
  defined as vaginal bleeding and / or uterine hypertonia, leading to emergency delivery, with evidence of retroplacental hematoma in the postpartum period. Yes / No categorical and dichotomous variable.
Maternal urinary tract infection | 1 month
  defined when urine culture is positive for any microorganism, and treatment has been started, regardless of symptoms. Yes / No categorical and dichotomous variable.
Maternal heart disease | 1 month
  presence of any congenital or acquired maternal heart disease, according to the patient's information, or diagnosed during hospitalization. Yes / No categorical and dichotomous variable.
Bronchial asthma | 1 month
  as reported by the patient and / or described in the medical record presenting the diagnosis of asthma. Yes / No categorical and dichotomous variable.
Chronic obstructive pulmonary disease (COPD) | 1 month
  as reported by the patient and / or described in the medical record presenting the diagnosis of COPD. Yes / No categorical and dichotomous variable.
Cerebrovascular disease | 1 month
  as reported by the patient and / or described in the chart that presents the diagnosis of cerebrovascular disease. Yes / No categorical and dichotomous variable.
Chronic kidney injury | 1 month
  as reported by the patient and / or described in the chart that presents the diagnosis of CRL. Yes / No categorical and dichotomous variable.
Immunosuppression | 1 month
  as reported by the patient and / or described in the chart that presents the diagnosis of immunosuppressive disease or use immunosuppressive medication. Categorical and dichotomous Yes / No type.
Maternal pneumonia | 1 month
  presence of the flu syndrome associated with laboratory changes, such as leukocytosis or leukopenia, and radiological, such as localized or diffuse interstitial infiltrate, or presence of a condensation area, as diagnosed by the attending physician. Yes / No categorical and dichotomous variable.
Maternal sepsis | 1 month
  life-threatening organ dysfunction resulting from an unregulated response by the body to an infection. Yes / No categorical and dichotomous variable.
Septic shock | 1 month
  defined as a situation of sepsis, associated with signs of hypoperfusion, with fluid-refractory hypotension and requiring vasopressor therapy (Lactate> 2 mmol / L). Yes / No categorical and dichotomous variable.
Severe acute respiratory syndrome (SARS) | 1 month
  flu-like syndrome (fever, cough, dyspnoea and other nonspecific), accompanied by oxygen saturation <95% (SatO2), respiratory distress or tachypnea, hypotension and worsening of the clinical conditions of the underlying disease. Yes / No categorical and dichotomous variable.
Postpartum hemorrhage | 14 days
  increased postpartum bleeding, according to the assessment of the attending physician, requiring some maneuver or therapy for control. Yes / No categorical and dichotomous variable.
Infection of the operative site | 14 days
  exit of purulent secretion by the surgical scar, according to the assessment of the attending physician. Yes / No categorical and dichotomous variable.
Endometritis | 14 days
  characterized by the discharge of purulent secretion from the uterine cervix, remaining dilated, with an unpleasant odor and fever for a minimum of two consecutive days, excluding the first 24 hours, according to the assessment of the attending physician. Yes / No categorical and dichotomous variable.
Peritonitis | 14 days
  characterized by abdominal pain, with compatible image examination, according to the assessment of the attending physician. Categorical and dichotomous Yes / No type.
Need for postpartum hysterectomy | 1 month
  removal of the uterus, for any indication, according to the assessment of the attending physician. Yes / No categorical and dichotomous variable.
Type of delivery | 1 hour
  defined as the type of delivery performed, categorized as normal, instrumental (vacuum or forceps) or cesarean delivery.
Indication of cesarean section | 1 hour
  if a cesarean section was performed, insert the indication that the attending physicians described, which can be later modified, according to the medical record evaluation by the researchers. The main indications are: dystocias, including cephalopelvic disproportion, macrosomia, impaired fetal vitality, placenta previa, cord prolapse, placental abruption, among others.
Gestational age at birth | 1 hour
  gestational age at birth, in weeks, calculated by the day of the last menstruation and confirmed by the first ultrasound scan of the amniocentesis. Numerical and discrete variable.
Use of labor analgesia | 4 hours
  use of pharmacological labor analgesia, as indicated by the attending physician and declared in medical records. Yes / No categorical and dichotomous variable.
Type of anesthesia for cesarean section | 1 hour
  method of anesthesia for performing cesarean section, categorized into spinal anesthesia, epidural and general anesthesia.
Antenatal corticosteroid therapy (pulmonary maturity) | 14 days
  as noted in the medical records, referring to the complete course of betamethasone (12mg two doses in a 24h interval) or dexamethasone (6mg 12 / 12h, for two days), incomplete course, not taking corticosteroids or without indication for accelerating fetal lung maturity.
Use of maternal magnesium sulphate (prophylaxis of the newborn and / or prevention of eclampsia) | 32 weeks
  as noted in the medical record, magnesium sulphate for neuroprotection, before delivery and until the 32nd week of pregnancy, being categorized as complete course (performance of attack and first stage of magnesium sulfate before delivery), incomplete, not performed or without indication.
Maternal prophylactic antibiotic therapy (prophylaxis of neonatal sepsis) | 14 days
  as noted in the medical records, referring to the use of the prophylactic regimen of crystalline penicillin to prevent neonatal infection with group B Streptococcus, being categorized as complete (completion of at least two phases) crystalline penicillin before delivery), incomplete, not performed or without indication.
Hospital discharge when pregnant | 1 month
  when the pregnant patient was admitted and discharged while pregnant. Yes / No categorical and dichotomous variable.
Hospital discharge when puerperal | 1 month
  when the pregnant or puerperal patient has been admitted and discharged in the puerperal state. Yes / No categorical and dichotomous variable.
Maternal death when pregnant | 1 month
  when maternal death occurs with the pregnant patient. Categorical and dichotomous Yes / No type.
Maternal death when puerperal | 45 days
  when maternal death occurs with the patient in the puerperal state. Categorical and dichotomous Yes / No type.
Fetal death | 10 hours
  birth of a fetus without vitality. Yes / No categorical and dichotomous variable.
Perinatal death | 27 days
  fetal or neonatal death (up to and including the 27th day of life). Yes / No categorical and dichotomous variable.
Birth weight | 1 hour
  as measured on a standard scale, in the delivery room, in grams, and recorded in medical records. Numerical and discrete variable.
Adequacy of birth weight | 1 hour
  classification of birth weight, according to gestational age, being categorized as: small for gestational age (SGA), when <10th pct; suitable for gestational age (AGA), when between 10º pct and 90º pct; and great for gestational age (GIG), when> 90º pct.
Apgar scores in the first minute | 1 minute
  as calculated by the classic Apgar score , in the first minute of birth, recorded in medical records, which can be later categorized. Numerical and discrete.
Apgar scores in the fifth minute | 5 minutes
  as calculated by the classic Apgar score, in the fifth minute of birth, recorded in medical records, which can be further categorized. Numerical and discrete variable.
Neonatal ICU admission | 1 hour
  defined as the newborn's stay in the neonatal intensive care unit after delivery, to perform any procedure. Yes / No categorical and dichotomous variable.
Need for neonatal resuscitation | 27 days
  defined as the need for resuscitation maneuvers, performed on the newborn, in the delivery room or until the 27th day after delivery. Yes / No categorical and dichotomous variable.
Need for neonatal mechanical ventilation | 27 days
  defined as the need for assisted mechanical ventilation, provided to the newborn, in the delivery room or until the 27th day after delivery. Yes / No categorical and dichotomous variable.
Neonatal nasal catheter | 27 days
  need for a neonatal nasal catheter to maintain normal oxygen saturation. Yes / No categorical and dichotomous variable.
Neonatal Continuous Positive Airway Pressure (CPAP) mask | 27 days
  need for neonatal CPAP to maintain normal oxygen saturation. Yes / No categorical and dichotomous variable.
Neonatal hypothermia | 27 days
  defined when the axillary temperature is less than or equal to 35ºC, as noted in the medical record for neonatal care. Yes / No categorical and dichotomous variable.
Neonatal hypoglycemia | 27 days
  defined as peripheral blood glucose below 40mg / dl, as noted in the medical record for neonatal care. Yes / No categorical and dichotomous variable.
Neonatal infection | 27 days
  defined as any neonatal infection diagnosed as noted in the medical record by neonatal care. Yes / No categorical and dichotomous variable.
Chorioamnionitis | 27 days
  defined as the infection of the amniotic cavity, as noted in the medical record for neonatal care. Yes / No categorical and dichotomous variable.
Neonatal respiratory distress modality | 1 month
  defined as newborn's respiratory distress (RDS), transient tachypnea of the newborn (NRT) or absent respiratory distress, as noted in the medical record for neonatal care.
Neonatal congenital infection (TORCHS) | 1 month
  defined as any congenital infection confirmed at birth, based on fetal PCR, neonatal examination or maternal serology, as noted in the medical record for neonatal care. Yes / No categorical and dichotomous variable.
Congenital malformation | 1 month
  defined as any fetal congenital malformation present, as noted in medical records by neonatal care. Yes / No categorical and dichotomous variable.
Breastfeeding | 1 month
  exclusive breastfeeding, during hospitalization, by natural method or pasteurized breast milk. Yes / No categorical and dichotomous variable.
Cord ligation | 10 minutes
  can be divided into early, when performed in less than three minutes, and timely, when between three to five minutes. Categorical and dichotomous variable.
Skin-to-skin contact | 1 hour
  as early contact was made between the mother and the baby, early, still in the delivery room. Yes / No categorical and dichotomous variable.
Breastfeeding in the delivery room | 1 hour
  according to breastfeeding, early, still in the delivery room. Yes / No categorical and dichotomous variable.
Days of life of the newborn's diagnostic suspicion | 1 month
  days of life of the newborn until the newborn's diagnostic suspicion. Numerical and discrete variable.
Result of the Polymerase Chain Reaction - Real Time (RT-PCR) for neonatal COVID-19 in diagnosis, at 6 months, 12 months and 24 months | 6 months, 12 months and 24 months
  result of RT-PCR in the diagnosis of COVID-19, through the blood or nasopharyngeal secretion, according to the usual technique, being categorized as positive, negative and indeterminate.
Result of Polymerase Chain Reaction - Real Time (RT-PCR) for the differential diagnosis of neonatal respiratory syndrome (viral panel) | 6 months, 12 months and 24 months
  result of RT-PCR in the differential diagnosis of respiratory syndrome, through blood or nasopharyngeal secretion, according to the technique and kit used, being categorized as positive (any virus found), negative and indeterminate.
Neonatal viral panel in the diagnosis, at 6 months, 12 months and 24 months | 6 months, 12 months and 24 months
  result of RT-PCR of the viral panel in the differential diagnosis of respiratory syndrome, through blood or nasopharyngeal secretion, according to the technique and kit used, categorized according to the virus found.
Neonatal cytokines | 6 months, 12 months and 24 months
  substances capable of modulating the cellular response of several cells, such as interleukins - IL-1ra, IL-6, IL-2, IL-5, IL-10, IL-12, IL-13, IL17A, IL -4, IL-1β, IL-9, IL-15, Interferon - IFN-γ and Tumor necrosis factor - TNF-α, in neonatal blood, in pg / ml, from the beginning of the flu syndrome or COVID-19 and in the period of the syndrome. Numeric and continuous variable (for each cytokine)
Neonatal IgM COVID-19 | 5 days
  result of IgM COVID-19 serology, using neonatal blood, according to the Enzyme-Linked Immunosorbent Assay (ELISA) technique or immunochromatography or chemiluminescent immunoassay, being categorized as positive, negative and indeterminate, according with the reference values of each serological kit, performed after the 5th day of signs and symptoms.
IgA COVID-19 neonatal serial | 5 days
  result of IgA COVID-19 serology, through neonatal blood, according to the ELISA technique, being categorized as positive, negative and indeterminate, according to the reference values of each serological kit, performed after the 5th day of signs and symptoms.
Serial neonatal IgG COVID-19 | 14 days
  result of IgG COVID-19 serology, through neonatal blood, according to the ELISA technique, being categorized as positive, negative and indeterminate, according to the reference values of each serological kit, performed after the 14th day of signs and symptoms. Numeric and continuous variable.
Neonatal reinfection | 14 days
  after diagnostic confirmation of COVID-19 and 14 days after the cure criteria, the RT-PCR test returns positive. Yes / No categorical and dichotomous variable.
Hemoglobin from neonatal diagnosis | 14 days
  value of the first hemoglobin measured in neonatal blood, in g / dL, from the suspicion of the diagnosis by COVID-19. Numeric and continuous variable.
Diagnostic neonatal bleeding time (BT) | 1 month
  value of the first BT measured in neonatal blood, in seconds (s), from the suspicion of the diagnosis by COVID-19. Numerical and discrete variable.
Diagnostic neonatal clotting time (CT) | 1 month
  value of the first CT measured in neonatal blood, in seconds (s), from the suspicion of the diagnosis by COVID-19. Numerical and discrete variable.
Urea from neonatal diagnosis | 1 month
  value of the first urea measured in neonatal blood, in mg / dL, from the suspicion of the diagnosis by COVID-19. Numerical and discrete variable.
Creatinine from neonatal diagnosis | 1 month
  value of the first creatinine measured in neonatal blood, in mg / dL, based on the suspected diagnosis by COVID-19. Numerical and discrete variable.
Transaminases of the neonatal diagnosis | 1 month
  defined as aspartate aminotransferase or glutamic-oxalacetic transaminase and alanine aminotransferase or glutamic-pyruvic transaminase, based on the suspicion of the diagnosis by COVID-19.
Blood culture of the neonatal diagnosis | 1 month
  result of the first blood culture, from the suspicion of the diagnosis by COVID-19, categorized as negative and positive (growth of the microorganism). Categorical and dichotomous variable.
Uroculture of neonatal diagnosis | 1 month
  result of the first urine culture, based on the suspicion of the diagnosis by COVID-19, categorized as negative and positive (growth of the microorganism). Categorical and dichotomous variable.
IgM COVID-19 - worst neonatal result | 5 days
  worst result of IgM COVID-19 serology, using neonatal blood, according to the Enzyme-Linked Immunosorbent Assay (ELISA) technique or immunochromatography or chemiluminescent immunoassay, being categorized as positive, negative and indeterminate , according to the reference values of each serological kit, performed after the 5th day of signs and symptoms.
Neonatal IgG COVID-19 - worst serial result | 14 days
  worst result of IgG COVID-19 serology, through blood, according to the ELISA technique, being categorized as positive, negative and indeterminate, according to the reference values of each serological kit , performed after the 14th day of signs and symptoms. Numeric and continuous variable.
Cytokines - worst neonatal result | 14 days
  worst result of cytokines, substances capable of modulating the cellular response of several cells, such as interleukins - IL-1ra, IL-6, IL-2, IL-5, IL-10, IL-12 , IL-13, IL17A, IL-4, IL-1β, IL-9, IL-15, Interferon - IFN-γ and Tumor necrosis factor - TNF-α, in neonatal blood, in pg / ml, from suspected diagnosis. Numeric and continuous variable (for each cytokine).
Day of the worst blood count result from the beginning of the suspected diagnosis by COVID-19 | 1 month
  day of the worst blood count result, from the suspicion of the diagnosis by COVID-19. Numerical and discrete variable.
Day of the worst value of the neonatal coagulogram from the suspicion of the diagnosis by COVID-19 | 1 month
  day of the realization of the worst value of the coagulogram, from the suspicion of the diagnosis by COVID-19. Numerical and discrete variable.
Bleeding time - worst neonatal result (BT) | 1 month
  value of the worst BT result measured in neonatal blood, in seconds (s), from the suspicion of the diagnosis by COVID-19. Numerical and discrete variable.
Urea - worst neonatal result | 1 month
  value of the worst result of urea measured in neonatal blood, in mg / dL, based on the suspicion of the diagnosis by COVID-19. Numerical and discrete variable.
Creatinine - worst neonatal result | 1 month
  value of the worst result of creatinine measured in neonatal blood, in mg / dL, based on the suspicion of the diagnosis by COVID-19. Numerical and discrete variable.
Transaminases - worst neonatal result | 1 month
  defined as the worst result of aspartate aminotransferase (AST) or glutamic oxalacetic transaminase and alanine aminotransferase or glutamic-pyruvic transaminase measurements, from the beginning of suspected COVID-19 diagnosis.
Blood culture - worst neonatal result | 1 month
  result of the worst blood culture, from the suspicion of the diagnosis by COVID-19, categorized as negative and positive (growth of the microorganism). Categorical and dichotomous variable.
Uroculture - worst neonatal result | 1 month
  result of the worst urine culture, from the suspicion of the diagnosis by COVID-19, categorized as negative and positive (growth of the microorganism). Categorical and dichotomous variable.
Gasometry - worst neonatal result | 1 hour
  defined as the worst result of measuring hydrogen potential, excess of bases, bicarbonate, partial pressure of oxygen (pO2), partial pressure of carbon dioxide (pCO2) and oxygenation index, in neonatal arterial blood, from the beginning of suspected COVID-19 diagnosis.
Result of RT-PCR of the placenta | 1 month
  result of RT-PCR in the diagnosis of COVID-19, through the placenta, according to the usual technique, being categorized as positive, negative and indeterminate.
Placental viral panel | 1 month
  result of the RT-PCR of the viral panel in the differential diagnosis of respiratory syndrome, through the placenta, according to the technique and kit used, categorized according to the virus found.
Histopathological of the placenta | 1 month
  result of the histopathological of the placenta, according to the usual technique.
Result of RT-PCR in breast milk at diagnosis, at birth and with and at hospital discharge | 1 month
  result of RT-PCR in the diagnosis of COVID-19, using breast milk, according to the usual technique, being categorized as positive, negative and indeterminate.
Viral panel in breast milk | 1 month
  result of RT-PCR of the viral panel in the differential diagnosis of respiratory syndrome, through breast milk, according to the technique and kit used, categorized according to the virus found.
Presence of alteration of the neonatal chest radiography | 1 day
  presence of any radiological alteration, described in a medical report. Yes / No categorical and dichotomous variable.
Result of neonatal chest radiography | 1 day
  description of any radiological changes, according to a medical report.
Presence of alteration of the neonatal chest tomography | 1 day
  presence of any alteration of the tomography, described in a medical report. Yes / No categorical and dichotomous variable.
Result of neonatal chest tomography | 1 day
  description of any alteration of the tomography, according to a medical report.
Parameters for monitoring the growth of the newborn at 6, 12 and 24 months - Head circumference | 6, 12 and 24 months
  measured by the assistant pediatrician as noted on the prenatal card, in grams. It can later be categorized, according to the WHO gestational age curve, 2006. Continuous numerical variable.
Parameters for monitoring the growth of the newborn at 6, 12 and 24 months - Weight | 6, 12 and 24 months
  measured by the assistant pediatrician as noted on the prenatal card, in grams. It can later be categorized, according to the WHO gestational age curve, 2006. Continuous numerical variable.
Parameters for monitoring the growth of the newborn at 6, 12 and 24 months - Height | 6, 12 and 24 months
  measured by the assistant pediatrician as noted on the prenatal card, in cm. It can later be categorized, according to the WHO gestational age curve, 2006. Continuous numerical variable.
Development of the newborn up to 6 months | 6 months
  as assessed by the responsible for the newborn and the assistant pediatrician and noted on the prenatal card. It will be considered as adequate, when all are present, and inappropriate, if any of the situations is absent: the baby is firmer and already sits with support; he turns around and rolls from side to side; grabs toys like rings and rattles, holding tight and resisting if someone tries to take them out of your hand; and when he hears some noise, he turns his head to find where it comes from.
Development of the newborn up to 12 months | 12 months
  as assessed by the responsible for the newborn and the assistant pediatrician and noted on the prenatal card. It will be considered as appropriate, when all are present, and inappropriate, if any of the situations is absent: the baby can stand up, leaning on furniture or with the help of a person; clap your hands, you can point with your finger what you want to catch and have fun saying goodbye; and you may be speaking a word or two like mom, pope, give.
Development of the newborn up to 24 months | 24 months
  as assessed by the responsible for the newborn and the assistant pediatrician and noted on the prenatal card. It will be considered as appropriate, when all are present, and inadequate, if any of the situations is absent: start to put two words together and speak simple phrases like "where's the cat?" or "milk not"; he demonstrates his own will, tests limits and speaks the word "no" a lot; climbs on chairs and sofas. Run, go up and down stairs, standing, with the help of an adult; can help to dress; and you can start to learn how to control pee and poop.

CONTACTS AND LOCATIONS:
Overall Officials: LEILA KATZ, MD, PhD, Principal Investigator — Instituto Materno Infantil Prof. Fernando Figueira
Locations (1):
- Instituto Materno Infantil Prof. Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Cunha CMP, Amorim MMR, Guendler JA, Souza ASR, Katz L. Clinical and epidemiological profile of pregnant and postpartum women affected by COVID-19 who required respiratory support. Rev Bras Ginecol Obstet. 2025 Apr 30;47:e-rbgo14. doi: 10.61622/rbgo/2025rbgo14. eCollection 2025. PMID 40406476